CLINICAL TRIAL: NCT02071810
Title: A Double-blind, Randomised, Placebo-controlled Study to Evaluate the Tolerability, Pharmacokinetics and Pharmacodynamics of Four Multiple Rising Dose Regimens of BIA 9-1067 in Healthy Male Volunteers
Brief Title: Tolerability, Pharmacokinetics and Pharmacodynamics of BIA 9-1067
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bial - Portela C S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BIA-91067-102
Record Dates: First submitted 2012-01-19; First posted 2014-02-26 (Estimated); Results first posted 2015-01-09 (Estimated); Last update posted 2015-12-24 (Estimated); Status verified 2015-11

CONDITIONS: Parkinson's Disease (PD)
Keywords: Parkinson's disease (PD); Opicapone; Bial; BIA 9-1067
MeSH Terms: conditions — Parkinson Disease | interventions — opicapone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- BIA 9-1067 5 mg (Experimental): BIA 9-1067 (OPC, Opicapone) 5 mg
  Interventions: Drug: BIA 9-1067
- BIA 9-1067 10 mg (Experimental): BIA 9-1067 (OPC, Opicapone) 10 mg
  Interventions: Drug: BIA 9-1067
- BIA 9-1067 20 mg (Experimental): BIA 9-1067 (OPC, Opicapone) 20 mg
  Interventions: Drug: BIA 9-1067
- BIA 9-1067 30 mg (Experimental): BIA 9-1067 (OPC, Opicapone) 30 mg
  Interventions: Drug: BIA 9-1067
- Placebo (Experimental): Placebo, PLC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIA 9-1067
  Other Names: OPC, Opicapone
  Arms: BIA 9-1067 10 mg; BIA 9-1067 20 mg; BIA 9-1067 30 mg; BIA 9-1067 5 mg
Drug: Placebo
  Other Names: PLC, Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the tolerability of BIA 9-1067 after multiple rising dose regimens of BIA 9-1067.

DETAILED DESCRIPTION:
Single centre, double-blind, randomised, placebo-controlled study of four dosage regimens of BIA 9-1067 in four groups of healthy male volunteers. In each group, the study will consist of an once-daily (o.d.) 8-day multiple-dose period. Progression to the next dose level will only occur if the previous dose level was considered to be safe and well tolerated. An appropriate interval (will separate the investigation of doses to permit a timely review and evaluation of safety data prior to proceeding to a higher dose level.

ELIGIBILITY:
Inclusion Criteria:

1. A signed and dated informed consent form before any study-specific screening procedure is performed.
2. Aged between 18 and 45 years, inclusive.
3. Healthy as determined by the investigator on the basis of medical history, physical examination, clinical laboratory test results, vital signs and digital 12-lead electrocardiogram (ECG).
4. Nonsmoker or smoker of fewer than 10 cigarettes per day as determined by history. Must be able to abstain from smoking during the inpatient stay.

Exclusion Criteria:

1. Any significant cardiovascular (e.g. hypertension), hepatic, renal, respiratory (e.g. childhood asthma), gastrointestinal, endocrine (e.g. diabetes, dyslipidemia), immunologic, dermatological, haematological, neurologic, or psychiatric disease.
2. Acute disease state (e.g., nausea, vomiting, fever, diarrhoea) within 7 days before study day 1.
3. History of drug abuse within 1 year before study day 1.
4. History of alcoholism within 1 year before day 1. Consumption of more than 50 g of ethanol per day (12.5 cL glass of 10° [10%] wine = 12 g; 4 cL of aperitif, 42° [42%] whiskey = 17 g; 25 cL glass of 3° [3%] beer = 7.5 g; 25 cL glass of 6° [6%] beer = 15 g
5. Have previously received BIA 9-1067.
6. Positive serologic findings for human immunodeficiency virus (HIV) antibodies, hepatitis B surface antigen (HBsAg), and/or hepatitis C virus (HCV) antibodies.
7. Positive findings of urine drug screen (eg, amphetamines, barbiturates, benzodiazepines, cannabinoids, cocaine, methadone, opiates, MDMA [3,4-methylenedioxy-methamphetamine; ecstasy]).
8. History of any clinically important drug allergy.
9. Prohibited Treatments: use of any investigational drug within 90 days or prescription drug within 30 days before investigational medical product (IMP) administration.
10. Consumption of any caffeine-containing products (e.g., coffee, tea, chocolate, or soda) in excess of 6 cups per day (or equivalent), of grapefruit, grapefruit-containing products, or alcoholic beverages within 24 before study day 1.
11. Use of any over-the-counter drugs including herbal supplements (except for the occasional use of acetaminophen [paracetamol], aspirin and vitamins ≤100% recommended daily allowance) within 7 days before IMP administration.
12. Donation of blood (ie 450 ml) within 90 days before study day 1.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2008-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dikran Mouradian, MD, Principal Investigator — Biotrial
Locations (1):
- BIOTRIAL, Rueil, Malmaison, France

RESULTS

PARTICIPANT FLOW:
Groups:
- BIA 9-1067 5 mg: BIA 9-1067 (OPC, Opicapone) 5 mg
  BIA 9-1067
- BIA 9-1067 10 mg: BIA 9-1067 (OPC, Opicapone) 10 mg
  BIA 9-1067
- BIA 9-1067 20 mg: BIA 9-1067 (OPC, Opicapone) 20 mg
  BIA 9-1067
- BIA 9-1067 30 mg: BIA 9-1067 (OPC, Opicapone) 30 mg
  BIA 9-1067
- Placebo: Placebo, PLC
  Placebo
Period: Overall Study
Arm/Group | BIA 9-1067 5 mg | BIA 9-1067 10 mg | BIA 9-1067 20 mg | BIA 9-1067 30 mg | Placebo
Started | 6 | 6 | 6 | 7 | 9
Completed | 6 | 6 | 6 | 6 | 8
Not Completed | 0 | 0 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIA 9-1067 5 mg | BIA 9-1067 10 mg | BIA 9-1067 20 mg | BIA 9-1067 30 mg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 9 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 6 | 6 | 6 | 7 | 9 | 34
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 7 | 9 | 34

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With at Least One Adverse Event
Time Frame: participants will be followed for the duration of hospital stay, an expected average of 6 weeks
Measure: Number; unit: Number of patients
Arm/Group | BIA 9-1067 5 mg | BIA 9-1067 10 mg | BIA 9-1067 20 mg | BIA 9-1067 30 mg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 7 | 9
Number of patients | 3 | 1 | 1 | 2 | 1

ADVERSE EVENTS:
Arm/Group | BIA 9-1067 5 mg | BIA 9-1067 10 mg | BIA 9-1067 20 mg | BIA 9-1067 30 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/7 | 1/9
Other Adverse Events (participants affected / at risk) | 3/6 | 1/6 | 1/6 | 2/7 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 9-1067 5 mg (N=6) | BIA 9-1067 10 mg (N=6) | BIA 9-1067 20 mg (N=6) | BIA 9-1067 30 mg (N=7) | Placebo (N=9)
Left hemiparesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BIA 9-1067 5 mg (N=6) | BIA 9-1067 10 mg (N=6) | BIA 9-1067 20 mg (N=6) | BIA 9-1067 30 mg (N=7) | Placebo (N=9)
Headache (Nervous system disorders) | 3 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0 | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other